CLINICAL TRIAL: NCT01154946
Title: A New Approach to Clinical Implication of Detrusor After-contraction (DAC)
Brief Title: Clinical Implication of DAC (Detrusor After-contraction)
Acronym: DAC
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Hospital, Seoul National University Hospital
Other Study IDs: DAC; H-0805-056-245
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Voiding Dysfunction
Keywords: detrusor after-contraction; urodynamic; LUTS; urinary bladder, overactive; bladder dysfunction
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- DAC group: patients who show detrusor after-contraction during voiding cystometrography (CMG)

SUMMARY:
The aims of this study are

* to confirm whether detrusor after-contraction (DAC) is a true contraction or not with a new approach
* and to understand clinical implication of DAC

DETAILED DESCRIPTION:
The definition of detrusor after-contraction (DAC) is usually accepted as the increase of detrusor pressure (Pdet), whether it is sudden or not, after cessation of urinary flow. The amount of increase in Pdet is sometimes included in the definition of DAC (14, 15, 20 cmH2O or at least two times the level of the maximal Pdet during the voiding phase). However, it is clear that the lack of a well-established definition may induce much bias in the interpretation of the clinical implication of DAC. The previous studies showed a wide range of prevalence.1-4 DAC seemed to occur more frequently in children and the occurrence rate usually decreased with age in urodynamic studies.

ELIGIBILITY:
Inclusion Criteria:

* Indications and selection of patients for conduction of urodynamic studies (UDS) were followed as the recommendation of ICS (international continence society).

Exclusion Criteria:

* Patients with indwelling catheters, urinary tract infection and urinary stones were excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2,309 patients more than 18 years old with neurogenic or non-neurogenic voiding dysfunction who performed urodynamic studies
Sampling Method: Non-Probability Sample
Enrollment: 2309 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to confirm whether DAC is a true contraction or not | up to 2 years (2007.Jan-2008.Dec)
  no change of Pdet when patients cough could confirm that DAC was a true contraction. Because an artifact occurred when a catheter was pressed against bladder wall or urethra, no change of intravesical pressure and increase of abdominal pressure finally induced a negative deflection of Pdet and this change of Pdet could be regarded as an artifact.

SECONDARY OUTCOMES:
Past medical history including neurological disorders and pelvic irradiation were also included in the database | up to 2 years (2007.Jan-2008.Dec)
  One-way analysis of variance and the chi-square test were performed to determine whether there was a relationship between the presence of DAC and the underlying neurogenic and non-neurogenic conditions

CONTACTS AND LOCATIONS:
Overall Officials: Seung-June Oh, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Ruarte AC, Podesta ML, Medel R. Detrusor after-contractions in children with normal urinary tracts. BJU Int. 2002 Aug;90(3):286-93. doi: 10.1046/j.1464-410x.2002.02827.x. PMID 12133067